CLINICAL TRIAL: NCT01339611
Title: Education Program for Patients Receiving Oral Anticoagulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Rosana Aparecida Spadoti Dantas, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OATeducation
Record Dates: First submitted 2011-04-13; First posted 2011-04-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2010-03

CONDITIONS: Cardiovascular Disease; Venous Thromboses; Atrial Fibrillation; Blood Coagulation Disorders, Inherited
Keywords: quality of life; medical adherence; warfarin; Health education
MeSH Terms: conditions — Cardiovascular Diseases; Venous Thrombosis; Atrial Fibrillation; Blood Coagulation Disorders, Inherited; Health Education

ARMS (2):
- Educational Program (Experimental): Patients who are going to use of oral anticoagulant will participate in an individual orientation, using instructional material (slides and illustrative booklet) during hospitalization period and the telephone follow-up at a week and four weeks after discharge
  Interventions: Behavioral: Educational program
- usual care (Other): Patients who are going to use of oral anticoagulant will have usual orientation from the health service (illustrative booklet) during hospitalization time. No telephone follow-up after discharge.
  Interventions: Behavioral: Educational program

INTERVENTIONS:
Behavioral: Educational program — Individual orientation (slides) during hospitalization period and telephone follow-up after discharge

SUMMARY:
The aim of the study is to test if patients under oral anticoagulation therapy who are going to participate in the education program will have better Health-related quality of life, higher rate in pharmacological treatment adherence and better self efficacy to manage the treatment.

DETAILED DESCRIPTION:
Patients who are going to use oral anticoagulant will participate in an individual orientation, using instructional material (slides and illustrative booklet) during hospitalization period. After the discharge 2 phone calls will be done (after: a week and four weeks) focusing on the strategies to improve patient's self-efficacy to manage the oral anticoagulation. There will be a personal contact among researcher and participants when the patients return at the oral anticoagulant ambulatory, two months after the treatment start. At this time the following variables of interest will be evaluated: Health-related quality of life; adherence to treatment and patients' self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in two public hospitals, in São Paulo state interior and who are going to start the use of oral anticoagulant during this hospitalization
* Patients admitted in two public hospitals, in São Paulo state interior and who are going to adjust therapeutically oral anticoagulant dosage or to start over treatment.

Exclusion Criteria:

* Individuals who do not at all have any ability to understand the data collection instrument questions, measured by the instrument Mental State Mini-exam.
* Individuals who do not have a telephone to be contacted after hospital discharge;
* Individuals who are going to metallic valve prosthesis implant surgery in the last six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in health-related quality of life at 2 months | baseline (hospitalization time) and two months after discahrge
  the health-related quality of life will be measure by Duke Anticoagulation Satisfaction Scale

SECONDARY OUTCOMES:
change from baseline in oral anticoagulation treatment adherence at 2 months | baseline (hospitalization time) and two months after discahrge
  Treatment adhrence will be measure by on specif scale

CONTACTS AND LOCATIONS:
Overall Officials: Flávia M Pelegrino, MNS, PhD candidate, Principal Investigator — University of São Paulo at Ribeirão Preto College of Nursing; Inaiara S.A. Corbi, MNS, PhD candidate, Principal Investigator — University of São Paulo at Ribeirão Preto College of Nursing; Rosana A.S. Dantas, PhD, Study Director — University of São Paulo at Ribeirão Preto College of Nursing
Locations (1):
- Hospital Estadual de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil